CLINICAL TRIAL: NCT01647802
Title: Cross-over Study of Three Modular Devices for Aid in Patient Standing and Transfer
Acronym: VTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: LOCAL/2012/EV-03; 2012-A00638-35 (Other: RCB number)
Record Dates: First submitted 2012-07-17; First posted 2012-07-24 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Mobility Limitation
Keywords: standing devices; transfer devices
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Turner-Vertic'Easy-Tina (Experimental): Standing will be attempted with the three devices in the following order: (1) Turner; (2) Vertic'Easy; (3) Tina.
  Interventions: Device: Standing attempts with the "Vertic'Easy" Device; Device: Standing attempts with the "Turner" Device; Device: Standing attempts with the "Tina" device
- Turner-Tina-Vertic'Easy (Experimental): Standing will be attempted with the three devices in the following order: (1) Turner; (2) Tina; (3) Vertic'Easy.
  Interventions: Device: Standing attempts with the "Vertic'Easy" Device; Device: Standing attempts with the "Turner" Device; Device: Standing attempts with the "Tina" device
- Vertic'Easy-Turner-Tina (Experimental): Standing will be attempted with the three devices in the following order: (1) Vertic'Easy; (2) Turner; (3) Tina.
  Interventions: Device: Standing attempts with the "Vertic'Easy" Device; Device: Standing attempts with the "Turner" Device; Device: Standing attempts with the "Tina" device
- Vertic'Easy-Tina-Turner (Experimental): Standing will be attempted with the three devices in the following order: (1) Vertic'Easy; (2) Tina; (3) Turner.
  Interventions: Device: Standing attempts with the "Vertic'Easy" Device; Device: Standing attempts with the "Turner" Device; Device: Standing attempts with the "Tina" device
- Tina-Turner-Vertic'Easy (Experimental): Standing will be attempted with the three devices in the following order: (1) Tina; (2) Turner; (3) Vertic'Easy.
  Interventions: Device: Standing attempts with the "Vertic'Easy" Device; Device: Standing attempts with the "Turner" Device; Device: Standing attempts with the "Tina" device
- Tina-Vertic'Easy-Turner (Experimental): Standing will be attempted with the three devices in the following order: (1) Tina; (2) Vertic'Easy; (3) Turner.
  Interventions: Device: Standing attempts with the "Vertic'Easy" Device; Device: Standing attempts with the "Turner" Device; Device: Standing attempts with the "Tina" device

INTERVENTIONS:
Device: Standing attempts with the "Vertic'Easy" Device — Included patients had never used any of the three devices evaluated in this study. Therefore the patient will make two attempts at standing on each device to enable him/her to get used to the device at the first attempt. A video recording will be made from a camera positioned laterally. Only the results of the second attempt will be a kinematic analysis and will be used for analyzes.
  Other Names: Vertic'Easy; Manufacturer : HMS-VILGO, Parc Eurasanté - 243, Rue Salvador Allendé 59120 LOOS LEZ LILLE,
Device: Standing attempts with the "Turner" Device — Included patients had never used any of the three devices evaluated in this study. Therefore the patient will make two attempts at standing on each device to enable him/her to get used to the device at the first attempt. A video recording will be made from a camera positioned laterally. Only the results of the second attempt will be a kinematic analysis and will be used for analyzes
  Other Names: Turner; Manufacturer : ETAC AB, Suède ; distributed in France by : FRANCE REHAB, ZA du Serroir, 54690 LAY SAINT CHRISTOPHE
Device: Standing attempts with the "Tina" device — Included patients had never used any of the three devices evaluated in this study. Therefore the patient will make two attempts at standing on each device to enable him/her to get used to the device at the first attempt. A video recording will be made from a camera positioned laterally. Only the results of the second attempt will be a kinematic analysis and will be used for analyzes
  Other Names: Tina; Manufacturer : ALTER ECO Santé, 9 Boulevard de Maurens, 31270 CUGNAUX

SUMMARY:
The main objective of this study is to evaluate via a physiological analysis of the movements involved in standing, the level of forward flexion of the spine (in cm on the horizontal axis) obtained with the apparatus "Tina" and to compare levels obtained in the same patients with stander/transfer devices "Turner" and "Vertic'Easy".

DETAILED DESCRIPTION:
Secondary objectives of this study are to compare the three devices in terms of:

* the level recovery of the spine on the vertical axis (vertical displacement C7, cm)
* standing time, defined by the time between the start of the forward flexion and the beginning of the vertical stabilization phase (seconds)
* the success rate of the verticalization of the patient (the attempt is considered successful when the vertical position is held for 10 seconds).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is in stable medical condition (no complications in the last 10 days)
* The patient is unable to stand up by his/her self and requires help during transfers
* The patient has muscular force (quadriceps) > 3 out of 5.

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a limited support from at least one lower limb
* The patient has an unstable fracture
* The patient has a fragile heart
* The patient has joint pain localized in the knee, hip or ankle.
* The patient has already used one of three mechanisms to help with standing and transfer used in this study
* Behavioral problems (opposition, agitation)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Level of forward flexion of the spine (position of maximum horizontal displacement of C7) | Baseline (Day 0; cross-sectional study)
  cm

SECONDARY OUTCOMES:
Level of standing (maximum vertical displacement C7) | Baseline (Day 0; transversal study)
  cm
Angle of hip flexion (angle formed by the line connecting the acromion and the greater trochanter with the line connecting the greater trochanter and the lateral femoral condyle) | Baseline (Day 0; transversal study)
  degrees
Standing time (time from start of forward flexion and the beginning of the vertical stabilization phase) | Baseline (Day 0; transversal study)
  seconds
Verticalization achieved (yes/no) | Baseline (Day 0; transversal study)
  yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Viollet, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France